CLINICAL TRIAL: NCT02619760
Title: ShorT and OPtimal Duration of Dual AntiPlatelet Therapy-2 Study
Acronym: STOPDAPT-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Takeshi Morimoto, Professor of Medicine, Kyoto University, Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1114; UMIN000019948 (Other: UMIN)
Record Dates: First submitted 2015-11-29; First posted 2015-12-02 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Coronary Artery Disease | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1-month DAPT (Active Comparator): 1-month dual antiplatelet therapy (DAPT) composed of aspirin and P2Y12 receptor antagonists , followed by 59-month clopidogrel monotherapy
  Interventions: Drug: 1-month DAPT
- 12-month DAPT (Active Comparator): 1-month dual antiplatelet therapy (DAPT) composed of aspirin and P2Y12 receptor antagonists with 11-month DAPT composed of aspirin and clopidogrel, followed by 48-month aspirin monotherapy
  Interventions: Drug: 12-month DAPT

INTERVENTIONS:
Drug: 1-month DAPT — 1-month dual antiplatelet therapy (DAPT) composed of aspirin and P2Y12 receptor antagonists
  Arms: 1-month DAPT
Drug: 12-month DAPT — 12-month dual antiplatelet therapy (DAPT) composed of aspirin and P2Y12 receptor antagonists
  Arms: 12-month DAPT

SUMMARY:
The purpose of this study is to evaluate the safety of reducing dual antiplatelet therapy (DAPT) duration to 1 month after implantation of the everolimus-eluting cobalt-chromium stent (CoCr-EES).

DETAILED DESCRIPTION:
The drug-eluting stents (DESs) are currently used in the majority of percutaneous coronary intervention (PCI) procedures. On the other hand, the problems of the first-generation DES (late adverse events, such as very late stent thrombosis) have been pointed out. Dual antiplatelet therapy (DAPT) has become a standard regimen after DES implantation and for fear of very late stent thrombosis, DAPT is frequently performed for 1 year or longer in clinical practice. However, serious hemorrhagic complications associated with a prolonged DAPT duration can bring disadvantages to patients, and it is extremely important to clarify an optimal DAPT duration after DES procedure. Currently, 1-month DAPT regimen after bare metal stent (BMS) implantation is commonly used in clinical practice, producing no major problems. Based on a meta-analysis of recent clinical studies, it has also been reported that the use of Cobalt-Chromium Everolimus-Eluting Stent (CoCr-EES) reduces the risk of early stent thrombosis by half compared to the use of BMS. There is no necessity to extend antiplatelet therapy after CoCr-EES implantation longer than after BMS implantation, and it is considered possible to use the same 1-month DAPT duration as after BMS implantation. The investigators therefore planned a multicenter, randomized, open-label, controlled study, in which the subjects who have undergone CoCr-EES procedure will be divided into the 1-month DAPT and clopidogrel monotherapy group and the 12-month DAPT and aspirin monotherapy group. Primary endpoint is the incidence of composite events including cardiovascular death, myocardial infarction, stent thrombosis, stroke, and bleeding defined by TIMI major or minor bleeding. At first, the non-inferiority about primary endpoint of 1-month DAPT group will be evaluated at 12 months after index procedure and secondarily, the superiority about primary endpoint of 1-month DAPT group will be evaluated at 5 years after index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients received percutaneous coronary intervention with cobalt-chromium everolimus-eluting stent
* Patients who are capable of oral dual antiplatelet therapy consisting of asprin and P2Y12 receptor antagonist

Exclusion Criteria:

* Patients requiring oral anticoagulants
* Patients with medical history of intracranial hemorrhage
* Patients who have experienced serious complications (myocardial infarction, stroke, and major bleeding) during hospital stay after percutaneous coronary intervention
* Patients with drug eluting stents other than Cobalt chromium everolimus eluting stents (Xience) implanted at the time of enrollment
* Patients comfirmed to have no tolerability to clopidgorel before enrollment
* Patients requiring continuous administration of antiplaelet drugs other than aspirin and P2Y12 receptor antagonists at the time of enrollment
* Patients with coronary bioabsorbable vascular scaffolds (BVS) implanted prior to or at the time of enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3045 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Composite event of cardiovascular death/myocardial infarction/definite stent thrombosis/stroke/bleeding | 12-month
  Composite event of cardiovascular death/myocardial infarction/definite stent thrombosis/stroke/bleeding defined as major or minor under the definition of Thrombolysis in Myocardial Infarction (TIMI) Study group

SECONDARY OUTCOMES:
Composite event of cardiovascular death/myocardial infarction/definite stent thrombosis/stroke | 12-month
Composite event of cardiovascular death/myocardial infarction/definite stent thrombosis/stroke | 60-month
Bleeding defined as major or minor under the definition of Thrombolysis in Myocardial Infarction (TIMI) Study group | 12-month
Bleeding defined as major or minor under the definition of Thrombolysis in Myocardial Infarction (TIMI) Study group | 60-month
Upper gastrointestinal endoscopic examination or treatment | 60-month
Composite event of all-cause death/myocardial infarction | 12-month
Composite event of all-cause death/myocardial infarction | 60-month
All-cause death | 12-month
All-cause death | 60-month
Composite event of cardiovascular death/myocardial infarction | 12-month
Composite event of cardiovascular death/myocardial infarction | 60-month
Cardiovascular death | 12-month
Cardiovascular death | 60-month
Myocardial infarction | 12-month
Myocardial infarction | 60-month
Stroke | 12-month
  a neurological deficit with acute onset that persists for at least 24 hours caused by a disturbance of the cerebral circulation due to ischemia or hemorrhage
Stroke | 60-month
  a neurological deficit with acute onset that persists for at least 24 hours caused by a disturbance of the cerebral circulation due to ischemia or hemorrhage
MACE (Major Adverse Cardiac Events) | 12-month
  Composite event of cardiac death, myocardial infarction and clinically-indicated target vesion revascularization
MACE (Major Adverse Cardiac Events) | 60-month
  Composite event of cardiac death, myocardial infarction and clinically-indicated target vesion revascularization
Definite stent thrombosis | 12-month
Definite stent thrombosis | 60-month
Target lesion failure | 12-month
  Composite event of cardiac death, myocardial infarction (MI) of target vessels, and Clinically-indicated TLR
Target lesion failure | 60-month
  Composite event of cardiac death, myocardial infarction (MI) of target vessels, and Clinically-indicated TLR
Target vessel failure | 12-month
Target vessel failure | 60-month
Target lesion revasucularization | 12-month
  PCI performed in the target lesion (within 5 mm of the stent edges), or CABG performed for restenosis of the target lesion or for treatment of other complications
Target lesion revasucularization | 60-month
  PCI performed in the target lesion (within 5 mm of the stent edges), or CABG performed for restenosis of the target lesion or for treatment of other complications
Clinically-driven target lesion revascularization | 12-month
  the revascularization that meets the following criteria; (1) recurrence of angina pectoris, presumably related to the target vessel, (2) objective signs of ischemia at rest or during exercise test (or equivalent), presumably related to the target vessel, (3) Signs of functional ischemia revealed by any invasive diagnostic test (e.g., Doppler flow velocity reserve [FVR], fractional flow reserve [FFR]), and (4) revascularization for ≥ 70% diameter stenosis even in the absence of the above-mentioned ischemic signs or symptoms. Presence/absence of clinical findings is judged by the operator of the procedure before the revascularization.
Clinically-driven target lesion revascularization | 60-month
  the revascularization that meets the following criteria; (1) recurrence of angina pectoris, presumably related to the target vessel, (2) objective signs of ischemia at rest or during exercise test (or equivalent), presumably related to the target vessel, (3) Signs of functional ischemia revealed by any invasive diagnostic test (e.g., Doppler flow velocity reserve [FVR], fractional flow reserve [FFR]), and (4) revascularization for ≥ 70% diameter stenosis even in the absence of the above-mentioned ischemic signs or symptoms. Presence/absence of clinical findings is judged by the operator of the procedure before the revascularization.
Non target lesion revascularization | 12-month
Non target lesion revascularization | 60-month
Coronary artery bypass graft | 12-month
Coronary artery bypass graft | 60-month
Target vessel revascularization | 12-month
Target vessel revascularization | 60-month
Any coronary reascluarization | 12-month
Any coronary reascluarization | 60-month
Bleeding complications | 12-month
  Evaluated with TIMI (major/minor/minimal), GUSTO (severe/moderate) and BARC (Type 1, 2, 3a, 3b, 3c, 4, 5a, 5b)
Bleeding complications | 60-month
  Evaluated with TIMI (major/minor/minimal), GUSTO (severe/moderate) and BARC (Type 1, 2, 3a, 3b, 3c, 4, 5a, 5b)
Gastrointestinal bleeding | 12-month
  Bleeding events requiring upper gastrointestinal endoscopic study or treatment.
Gastrointestinal bleeding | 60-month
  Bleeding events requiring upper gastrointestinal endoscopic study or treatment.
Gastrointestinal complaints | 12-month
  Symptoms requiring upper gastrointestinal endoscopic study or treatment
Gastrointestinal complaints | 60-month
  Symptoms requiring upper gastrointestinal endoscopic study or treatment
Newly diagnosed cancer | 60-month
  The endpoint is a newly diagnosed malignancy during the follow-up period that has not been previously diagnosed before enrollment. This does not include recurrent tumor after remission, includes early-stage cancer eligible for endoscopic treatment, and includes the tumors which are not diagnosed by tissue biopsy but are judged to be clinically malignant on imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, PhD, Study Chair — Professor of Medicine, Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Division of Cardiology, Kyoto University Hospital, Kyoto, Japan

REFERENCES:
- [Derived] Yamamoto K, Watanabe H, Morimoto T, Obayashi Y, Natsuaki M, Yamaji K, Domei T, Ogita M, Ohya M, Tatsushima S, Suzuki H, Tada T, Ishii M, Nikaido A, Watanabe N, Fujii S, Mori H, Nishikura T, Suematsu N, Hayashi F, Komiyama K, Shigematsu T, Isawa T, Suwa S, Ando K, Kimura T; STOPDAPT-2 and STOPDAPT-2 ACS Investigators. Clopidogrel Monotherapy After 1-Month Dual Antiplatelet Therapy in Patients With Diabetes Undergoing Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2023 Jan 9;16(1):19-31. doi: 10.1016/j.jcin.2022.09.053. Epub 2022 Dec 14. PMID 36599584
- [Derived] Obayashi Y, Watanabe H, Morimoto T, Yamamoto K, Natsuaki M, Domei T, Yamaji K, Suwa S, Isawa T, Watanabe H, Yoshida R, Sakamoto H, Akao M, Hata Y, Morishima I, Tokuyama H, Yagi M, Suzuki H, Wakabayashi K, Suematsu N, Inada T, Tamura T, Okayama H, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Morino Y, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 and STOPDAPT-2 ACS Investigators. Clopidogrel Monotherapy After 1-Month Dual Antiplatelet Therapy in Percutaneous Coronary Intervention: From the STOPDAPT-2 Total Cohort. Circ Cardiovasc Interv. 2022 Aug;15(8):e012004. doi: 10.1161/CIRCINTERVENTIONS.122.012004. Epub 2022 Aug 1. PMID 35912647
- [Derived] Watanabe H, Morimoto T, Natsuaki M, Yamamoto K, Obayashi Y, Ogita M, Suwa S, Isawa T, Domei T, Yamaji K, Tatsushima S, Watanabe H, Ohya M, Tokuyama H, Tada T, Sakamoto H, Mori H, Suzuki H, Nishikura T, Wakabayashi K, Hibi K, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Morino Y, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 ACS Investigators. Comparison of Clopidogrel Monotherapy After 1 to 2 Months of Dual Antiplatelet Therapy With 12 Months of Dual Antiplatelet Therapy in Patients With Acute Coronary Syndrome: The STOPDAPT-2 ACS Randomized Clinical Trial. JAMA Cardiol. 2022 Apr 1;7(4):407-417. doi: 10.1001/jamacardio.2021.5244. PMID 35234821
- [Derived] Yamamoto K, Watanabe H, Morimoto T, Domei T, Ohya M, Ogita M, Takagi K, Suzuki H, Nikaido A, Ishii M, Fujii S, Natsuaki M, Yasuda S, Kaneko T, Tamura T, Tamura T, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Igarashi Hanaoka K, Morino Y, Kozuma K, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 Investigators. Very Short Dual Antiplatelet Therapy After Drug-Eluting Stent Implantation in Patients Who Underwent Complex Percutaneous Coronary Intervention: Insight From the STOPDAPT-2 Trial. Circ Cardiovasc Interv. 2021 May;14(5):e010384. doi: 10.1161/CIRCINTERVENTIONS.120.010384. Epub 2021 May 18. PMID 34003662
- [Derived] Watanabe H, Morimoto T, Ogita M, Suwa S, Natsuaki M, Suematsu N, Koeda Y, Morino Y, Nikaido A, Hata Y, Doi M, Hibi K, Kimura K, Yoda S, Kaneko T, Nishida K, Kawai K, Yamaguchi K, Wakatsuki T, Tonoike N, Yamamoto M, Shimizu S, Shimohama T, Ako J, Kimura T; STOPDAPT-2 Investigators. Influence of CYP2C19 genotypes for the effect of 1-month dual antiplatelet therapy followed by clopidogrel monotherapy relative to 12-month dual antiplatelet therapy on clinical outcomes after percutaneous coronary intervention: a genetic substudy from the STOPDAPT-2. Cardiovasc Interv Ther. 2021 Oct;36(4):403-415. doi: 10.1007/s12928-020-00719-6. Epub 2020 Nov 12. PMID 33184726
- [Derived] Watanabe H, Domei T, Morimoto T, Natsuaki M, Shiomi H, Toyota T, Ohya M, Suwa S, Takagi K, Nanasato M, Hata Y, Yagi M, Suematsu N, Yokomatsu T, Takamisawa I, Doi M, Noda T, Okayama H, Seino Y, Tada T, Sakamoto H, Hibi K, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Hanaoka KI, Morino Y, Kozuma K, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 investigators. Details on the effect of very short dual antiplatelet therapy after drug-eluting stent implantation in patients with high bleeding risk: insight from the STOPDAPT-2 trial. Cardiovasc Interv Ther. 2021 Jan;36(1):91-103. doi: 10.1007/s12928-020-00651-9. Epub 2020 Feb 21. PMID 32086787
- [Derived] Watanabe H, Domei T, Morimoto T, Natsuaki M, Shiomi H, Toyota T, Ohya M, Suwa S, Takagi K, Nanasato M, Hata Y, Yagi M, Suematsu N, Yokomatsu T, Takamisawa I, Doi M, Noda T, Okayama H, Seino Y, Tada T, Sakamoto H, Hibi K, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Hanaoka KI, Morino Y, Kozuma K, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 Investigators. Effect of 1-Month Dual Antiplatelet Therapy Followed by Clopidogrel vs 12-Month Dual Antiplatelet Therapy on Cardiovascular and Bleeding Events in Patients Receiving PCI: The STOPDAPT-2 Randomized Clinical Trial. JAMA. 2019 Jun 25;321(24):2414-2427. doi: 10.1001/jama.2019.8145. PMID 31237644